CLINICAL TRIAL: NCT01026701
Title: Observational Study of Osteoblast Activity in Velcade�(Bortezomib) IV Treated Multiple Myeloma Patients.
Brief Title: Observational Study of the Effects Intravenous Bortezomib Has on Osteoblast (Cell That is Responsible for Bone Formation) Activity in Multiple Myeloma Patients.
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015067; 26866138MMY4036; BORKOR5020
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Myeloma
Keywords: Osteoblst effect; Velcade; Proteasome inhibitor; Bortezomib; Multjple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 001: bortezomib injection into a vein 1.3 mg/m2 twice a week for 21 days
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — injection into a vein 1.3 mg/m2 twice a week for 21 days

SUMMARY:
The purpose of this study is to measure the markers related to bone metabolism before and after the use of bortezomib injection in patients with multiple myeloma and to evaluate the effect bortezomib injection has on bone disease.

DETAILED DESCRIPTION:
Among several symptoms in patients with multiple myeloma, the bone disease is one of the most common symptoms that approximately 80 percent of the patients experience. Multiple myeloma is different from other tumors in that several osteoclast activating factors (OAF) released from multiple myeloma cells resorb bone and, at the same time, activation of osteoblast is inhibited, leading to unbalance of breakdown and formation of bone. Activation of osteoclast and inhibition of osteoblast brings about bone fractures, osteoporosis, hypercalcemia, bone pain and spinal cord compression. Those symptoms are directly related to patients' quality of life. Therefore, they are the important therapeutic targets for multiple myeloma. Various types of bisphosphonate agents are used for the treatment of the bone disease in patients with multiple myeloma. This is a prospective (a study where the participants are identified and then followed forward in time), multi-center, Phase 4, observational study (studies that record specific events occurring without any intervention from the researcher) in order to analyze the change in bone metabolism markers (DKK-1, sRANKL, OPG, sRANKL/OPG,bALP, OC) before and after the use of bortezomib injection by using an enzyme-linked immunosorbent assay (ELISA) in serum. The adverse events will be assessed through the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE V3). The patients will receive bortezomib injection into a vein 1.3 mg/m2 twice a week for 21 days under usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Among patients who are newly prescribed bortezomib injection as a secondary agent for the treatment of multiple myeloma, those of whom agree to provide information will be included.

Exclusion Criteria:

* Patients who are hypersensitive to the study drug or any component of the study drug or with a history of the hypersensitivity
* Patients with severe hepatic impairment
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who are newly prescribed bortezomib injection as a secondary agent for the treatment of multiple myeloma, those of whom agree to provide information will be included in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
bone metabolism markers (DKK-1, sRANKL, OPG, sRANKL/OPG,bALP, OC) | on day 1 at the first cycle, and 12-24 weeks

SECONDARY OUTCOMES:
CR rate | at the end of every 3 week cycle
Overall response rate | at the end of every 3 week cyclet
Correlation between primary endpoints and response rate | 12 -24 weeks
NRS pain score | at the end of every 3 week cycle
Adverse events | at the end of every 3 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.